CLINICAL TRIAL: NCT01585012
Title: Phase 2 Human Factors Usability Study of the Focus Touch™ Conception System: Semen Collection
Brief Title: Usability Study of the Focus Touch™ Conception System: Semen Collection
Acronym: Ib2C
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rinovum Women's Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 11-045
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Infertility
Keywords: Cervical cap insemination; Collection condom; Instructions for Use; Safety during intercourse; Acceptability of the cervical cap with condom sheath; slip; break; ease of conversion; adequate sample collection
MeSH Terms: conditions — Infertility | interventions — Contraceptive Devices, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cervical cap (Experimental): Collection condom with cervical cap inserted
  Interventions: Device: Cervical cap (Focus Touch™ Conception System)

INTERVENTIONS:
Device: Cervical cap (Focus Touch™ Conception System) — Cervical cap

SUMMARY:
This is a human factors usability study designed to validated usability by obtaining feedback in a home use environment regarding ease of use of the Focus Touch™ Conception System Conceptacle (when used to collect semen) and the instructions for use. The investigators will collect data to demonstrate that the usability requirements of the conception system as collection device, as determined by Usability Specification: Focus Touch Conception System, ER-000001 have been met. The ability of the device to be used during sexual intercourse without discomfort or injury to the female participant's vaginal/cervical tissues shall also be taken into account. Participating couples will be asked to use the Focus Touch™ Conception System Conceptacle (in condom form), using the Instructions For Use, to collect semen during sexual intercourse in a home use environment. This study will involve sexual intercourse between monogamous, heterosexual couples who are trying to conceive or are on a non-vaginal birth control with which they do not normally use condoms. Participants will be asked to complete the study and the questionnaire within 3 days of receiving the study packet. Contact information shall be collected, but participants will only be contacted if they fail to return the questionnaire within the requested timeframe.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual, monogamous couples, of any race or ethnicity, who are sexually active
* 20 - 50 years of age
* Signed Informed Consent
* Past experience with using condoms
* Trying to conceive or using a non-vaginal birth control with which they do not normally use a condom.

Exclusion Criteria:

* Vaginal tract medical interventions with the last three (3) month
* Vaginal prolapse
* Full Hysterectomy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine if the Focus Touch™ Conception System Conceptacle is functionally acceptable and meets the user's needs and expectations when used in the home during sexual intercourse as a semen collection device. | 4 days
  Participating couples will be given the Focus Touch™ Conception System Conceptacle. The Conceptacle will be used during sexual intercourse, in the home, to collect semen. The device will be used in accordance with the instructions for use. Participants will be asked to complete the study and the questionnaire within 3 days of receiving the study packet. Contact information shall be collected, but participants will only be contacted if they fail to return the questionnaire within the requested timeframe. As a result, this study could take up to 4 days to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Pelekanos, OB-GYN, Principal Investigator — Forbes Regional
Locations (1):
- Forbes Regional Hospital, Monroeville, Pennsylvania, United States